CLINICAL TRIAL: NCT03651297
Title: Testing a Simple Fall-arrest Harness vs. an Actuated and Instrumented Harness in Balance Training
Brief Title: Simple Fall-Arrest Harness vs. Adjustable Harness
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lab closed due to Covid 19
Sponsor: Cleveland State University (Other)
Responsible Party: Principal Investigator, Debbie Espy, Associate Professor, Cleveland State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2018-324
Record Dates: First submitted 2018-08-14; First posted 2018-08-29 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Fall Accident; Fall Injury; Balancing Interference
Keywords: Harness Assist; Balance training; Types of harness assist; Fall-arrest harness; Adjustable harness

STUDY DESIGN:
Intervention Model Description: The first group will complete two sessions of harnessed video gaming balance training. The second group will include older adults over the age of 50 with self-reported falls or the fear of falling. The second group of older adults will complete two sessions of a reactive (slip) training protocol. For both groups, the first session participants will be assigned randomly to use a standard fall-arrest harness or the new BWS harness system. At the second session, they will switch the harness used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Younger Adults (Experimental): First group will include 20 young adults with no history of falls or fear of falling. They will complete both interventions: Balance Training with Fall-Arrest Harness and Balance Training with Adjustable Harness.
  Interventions: Other: Balance training with Fall-Arrest harness; Other: Balance training with Adjustable harness
- Older adults (Experimental): Second group will include 20 older adults with a self-reported history of falls or fear of falling. They will complete both interventions: Balance Training with Fall-Arrest Harness and Balance Training with Adjustable Harness.
  Interventions: Other: Balance training with Fall-Arrest harness; Other: Balance training with Adjustable harness

INTERVENTIONS:
Other: Balance training with Fall-Arrest harness — This study will analyze the subjects' responses to balance training protocols with two types of harness support. The protocol will involve balance training, initially of low intensity and then advanced by an algorithm based on subjects' responses to the prior repetition of balance activity. For this intervention, the subjects will be using a standard Fall-Arrest harness for safety throughout, but no other external support. This will allow comparison of postural control, slip responses, motor learning, reliance on the harness and confidence with the system between the two harness types.
Other: Balance training with Adjustable harness — This study will analyze the subjects' responses to balance training protocols with two types of harness support. The protocol will involve balance training, initially of low intensity and then advanced by an algorithm based on subjects' responses to the prior repetition of balance activity. For this intervention, the subjects will be using a motorized harness in which the support provided is adjustable. This will allow comparison of postural control, slip responses, motor learning, reliance on the harness and confidence with the system between the two harness types.

SUMMARY:
Fall risk increases with age and the fear of falling can significantly impact activity, mobility and future fall risk. Exercise designed specifically to help balance is effective at improving balance and postural control for mobility, gait, and other daily activities. The individual purposes of this research are to (1) effectively use a prototype of an instrumented and actuated harness and support system, (2) demonstrate that this system can be used as designed during induced falls (reactive) and in place gaming (proactive) balance training protocols with the ability to modulate parameters as designed, measurements of harness system are accurate, and resultant output of the system matches intended parameters, and (3) demonstrate that the use of this system can allow provision of and study of varied balance training protocols, including: the measurements of the system, feedback of the system to participants, and the impact of the support parameters of the harness system on the task execution, learning and transfer.

Two separate groups of 20 participants (40 total participants) will be studied. The first group will include 20 individuals between the ages of 18 to 40 years old with no history of falls or fear of falling. The first group will complete two sessions of harnessed video gaming balance training. The second group will include older adults over the age of 55 with self-reported falls or the fear of falling. The second group of older adults will complete two sessions of a reactive (slip) training protocol. For both groups, the first session participants will be randomly assigned to use either a standard fall-arrest harness or the new BWS harness system. At the second session, they will switch the harness used. The protocol will involve slips or gaming based balance training, initially of low intensity and then advanced by algorithm based on their response to the trial just prior. This will allow comparison of postural control, perturbation responses, motor learning, and confidence with the system between the two harness types.

DETAILED DESCRIPTION:
Fall risk increases with age and the fear of falling can significantly impact activity, mobility and future fall risk. Exercise designed specifically to help balance is effective at improving balance and postural control for mobility, gait, and other daily activities. Balance training for fall prevention can be proactive or reactive. Proactive balance training is the practice of anticipatory and self-initiated movement. Reactive training, on the other hand, involves responses to unexpected movements that cause a loss of balance. Safety harness systems are used for reactive balance protocols to prevent actual falls. They may also be used in intense proactive protocols for more vulnerable, frail, or fearful participants. In therapeutic settings, harnesses for gait and mobility training are either body weight supporting (BWS) or fall-arresting.

The investigators have designed and built a harness system that allows better control of more of the support parameters than much more expensive, commercially available, and BWS systems. This harness system better controls aspects such as: limiting fall distance, modulation of how the support responds to descents, assist to return to stand, and recording of all body movements. This will allow the investigation of questions about the impact of harness systems on learning and performance of postural control and effective use of harnesses in balance training.

The investigators have done extensive work with the Xbox system using Kinect, having designed a protocol and progression of games and surfaces that provides high intensity proactive balance training using Kinect. The investigators also train reactive balance through the use of a custom made platform called the Slip Trainer (MASS Rehab, Dayton, OH), along with a fall arresting harness and load measuring device. This allows the administration of repeated slip perturbations of a consistent and known intensity safely and efficiently.

Questions that still need to be answered include: Will patients challenge themselves more or engage in more intense activities with a harness? Does the support provided by a harness impact or interfere with the motor learning of the balance tasks? Could balance task learning be more effective with some degree of support vs. just a fall-arresting "backup" as is theorized with treadmill gait training? If so, what types and parameters are most effective? Would this type of support allow more intense training to be extended to people who are less mobile, more vulnerable or frail or more fearful, those who would not be able to participate in effective balance training otherwise?

This study will answer initial questions about the effectiveness and acceptance of the harness system by older adults in a reactive and by younger adults in a proactive protocol, and will provide pilot data for larger, external grants to investigate the broader questions among a much larger group of people. The larger impact will be translating the technology and understanding its impact clinically, allowing much greater intensity and more effective balance training for at risk populations.

The investigators propose to build a harness system in which the support within a single plane can be finely controlled and measured. This harness will have the following capabilities: limit height/fall to a pre-set vertical limit with ability to modulate the fall arrest kinematics, dynamic partial body weight support - to remain constant with center of mass (COM) movements, modulate by pre-set thresholds how the support responds to descent, assist to return to stand - with preset thresholds and levels of assist, monitor/measure/record: vertical and horizontal components of body COM movements, and provide feedback to users re: the support of being provided or re: other parameters, potentially in various modes (haptic, visual, auditory).

The individual purposes of this research are to (1) effectively use a prototype of an instrumented and actuated harness and support system, (2) demonstrate that this system can be used as designed during induced falls (reactive) and in place gaming (proactive) balance training protocols with the ability to modulate parameters as designed, measurements of harness system are accurate, and resultant output of the system matches intended parameters, and (3) demonstrate that the use of this system can allow provision of and study of varied balance training protocols, including: the measurements of the system, feedback of the system to participants, and the impact of the support parameters of the harness system on the task execution, learning and transfer.

Two separate groups of 20 participants (40 total participants) will be studied. Participants will be recruited from students, faculty and staff, as well as community members known to the investigator following the procedure outlined below. The first group will include 20 individuals between the ages of 18 to 40 years old with no history of falls or fear of falling. The first group will complete two sessions of harnessed video gaming balance training. The second group will include older adults over the age of 55 with self-reported falls or the fear of falling. The second group of older adults will complete two sessions of a reactive (slip) training protocol. For both groups, the first session participants will be randomly assigned to use a standard fall-arrest harness or the new BWS harness system. BWS harness can be set to support a predetermined portion of the person's body weight and maintain that support throughout the session. At the second session, they will switch the harness used. The protocol will involve balance training, advanced by algorithm, based on the participant's response to the trial just prior. This will allow comparison of postural control, perturbation responses, motor learning, and confidence with the system between the two harness types.

ELIGIBILITY:
Inclusion Criteria:

* Age
* Completed Informed Consent
* Self-reported risk or fear of falling

Exclusion Criteria:

* Medical Condition - they are not eligible if they self-identify as having any musculoskeletal, neuromuscular, cardiopulmonary, or other conditions that would limit them from participation.
* Allergic to adhesive tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change (improvement) in response to increasingly difficult perturbations, as measured by the Rate of Perceived Stability Score (RPS). | 2 sessions of 60 - 90 minutes, more than 3 days but less than three weeks apart.
  The protocols are advanced by algorithm. The reactive algorithm sets initial slip distance and force by the individual's leg length, weight, and MiniBEST (balance evaluation systems test). The result of each slip (harness loading and recovery steps) dictates the next condition as set forth in the algorithm. The proactive algorithm is a hierarchy of game and balance surface difficulty: participants begin at the same level and progress based on their Rate of Perceived Stability (RPS) score for each condition. The RPS self-rates balance task difficulty from 1 to 10 (least to most challenging). Advancing through more steps/more quickly with one harness indicates greater efficacy of that harness in balance skill acquisition. Because balance ability and the learning curve for balance tasks are highly individual, the outcome of interest is individual improvement in response to increasingly difficult perturbations, rather than standardized measure of balance ability across subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Espy, Principal Investigator — Cleveland State University
Locations (1):
- Cleveland State University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No